CLINICAL TRIAL: NCT00413998
Title: Randomized Evaluation of Mitral Annuloplasty During Coronary Artery Bypass Grafting for Moderate Functional Ischaemic Mitral Regurgitation.
Brief Title: Randomised Ischaemic Mitral Evaluation (RIME) Trial
Acronym: RIME
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Department of Health, United Kingdom (Other Government); British Heart Foundation (Other); British Medical Association (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); University Hospitals, Leicester (Other); Medical University of Silesia (Other); University Hospitals Bristol and Weston NHS Foundation Trust (Other); Blackpool Victoria Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2006HS020B; NIHR Portfolio ID 4129 (Other Grant/Funding Number: National Institute for Health Research)
Record Dates: First submitted 2006-12-19; First posted 2006-12-20 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Mitral Regurgitation; Coronary Artery Disease
Keywords: Functional ischaemic mitral regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency; Coronary Artery Disease | interventions — Mitral Valve Annuloplasty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CABG + Mitral valve repair (Experimental)
  Interventions: Procedure: CABG + Mitral valve annuloplasty
- CABG only (Active Comparator)
  Interventions: Procedure: CABG

INTERVENTIONS:
Procedure: CABG + Mitral valve annuloplasty — Patients will receive a mitral annuloplasty ring in addition to coronary artery bypass grafting.
  Arms: CABG + Mitral valve repair
Procedure: CABG — Patients will undergo coronary artery bypass grafting alone.
  Arms: CABG only

SUMMARY:
The study is a randomised controlled trial comparing two treatment strategies for patients with moderate functional ischaemic mitral regurgitation undergoing coronary artery bypass grafting (CABG). Patients will be randomised to receive either CABG alone or CABG plus mitral annuloplasty. The objective of the study is to determine if mitral annuloplasty in addition to CABG improves outcome in patients with moderate functional ischaemic mitral regurgitation.

DETAILED DESCRIPTION:
70 patients with moderate functional ischaemic MR who are undergoing CABG will be recruited. Patients will be randomised to undergo either CABG alone or CABG combined with mitral annuloplasty. Patients will be investigated at baseline, 3 months and 1 year after surgery to determine functional capacity, quality of life, and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing CABG.
2. Patients with moderate functional ischaemic mitral regurgitation without leaflet prolapse.

Exclusion Criteria:

1. Patients with severe LV dysfunction (EF less than 30%).
2. Patients with associated significant aortic valve disease.
3. Patients with significant co-morbidities: renal impairment (creatinine > 160), liver impairment (INR > 2.0, bilirubin > 40), or underlying chronic obstructive lung disease (FEV1:FVC ratio < 0.6).
4. Patients with NYHA class IV symptoms, unstable angina, acute pulmonary oedema or cardiogenic shock.
5. Patients unsuitable for surgery e.g. patients with advanced malignancy, unable to give informed consent.
6. Patients with structural abnormalities of the mitral valve e.g. papillary muscle rupture, chordal rupture, etc.
7. Patients with associated conditions which would significantly increase the risk of surgery.
8. Patients who have had previous cardiac surgery.
9. Patients with a previous history of endocarditis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2007-01; Primary Completion 2012-04 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Functional capacity | 1 year

SECONDARY OUTCOMES:
Left ventricular volumes | 1 year
Mitral regurgitation grade | 1 year
Neurohormonal levels | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: John R Pepper, MChir, FRCS, Study Chair — Royal Brompton & Harefield NHS Foundation Trust; Marcus Flather, MBBS, FRCP, Principal Investigator — Royal Brompton Hospital NHS Trust, London; K. M. John Chan, FRCS CTh, Principal Investigator — Royal Brompton Hospital NHS Trust, London
Locations (9):
- 1st Dept of Cardiothoracic Surgery, Medical University of Silesia, Katowice, Poland
- United Kingdom (8):
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Bristol Heart Institute, Bristol
  - Harefield Hospital, Harefield
  - Glenfield Hospital, Leicester, Leicester
  - Royal Brompton Hospital, London
  - Hammersmith Hospital, London
  - Heart Hospital, University College Hospital, London
  - St. Mary's Hospital, London

REFERENCES:
- [Background] Chan KM, Amirak E, Zakkar M, Flather M, Pepper JR, Punjabi PP. Ischemic mitral regurgitation: in search of the best treatment for a common condition. Prog Cardiovasc Dis. 2009 May-Jun;51(6):460-71. doi: 10.1016/j.pcad.2008.08.006. PMID 19410679
- [Background] Chan KM, Wage R, Symmonds K, Rahman-Haley S, Mohiaddin RH, Firmin DN, Pepper JR, Pennell DJ, Kilner PJ. Towards comprehensive assessment of mitral regurgitation using cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2008 Dec 22;10(1):61. doi: 10.1186/1532-429X-10-61. PMID 19102740
- [Result] Chan KM, Punjabi PP, Flather M, Wage R, Symmonds K, Roussin I, Rahman-Haley S, Pennell DJ, Kilner PJ, Dreyfus GD, Pepper JR; RIME Investigators. Coronary artery bypass surgery with or without mitral valve annuloplasty in moderate functional ischemic mitral regurgitation: final results of the Randomized Ischemic Mitral Evaluation (RIME) trial. Circulation. 2012 Nov 20;126(21):2502-10. doi: 10.1161/CIRCULATIONAHA.112.143818. Epub 2012 Nov 7. PMID 23136163